CLINICAL TRIAL: NCT03685799
Title: Impact of Histologic Concordance Between Biopsies and the Endoscopic Resection Specimen, in the Treatment of Barrett's Esophagus in Dysplasia, on the Recurrence of Dysplasia
Acronym: PatheBarett
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: PatheBarett-IPC 2016-005
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-09

CONDITIONS: Barretts Esophagus With Dysplasia
Keywords: Barretts Esophagus; Dysplasia
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DHG on Barrett's esophagus: patients with DHG on Barrett's esophagus on endoscopic biopsies followed by endoscopic resection
  Interventions: Diagnostic Test: Pathological revision

INTERVENTIONS:
Diagnostic Test: Pathological revision — Pathological revision

SUMMARY:
Influence of histological concordance on the risk of recurrence:

the histological concordance being the comparison between the biopsies and the endoscopic resection piece and its concordant response rate.

DETAILED DESCRIPTION:
Influence of histological concordance on the risk of recurrence:

the histological concordance being the comparison between the biopsies and the endoscopic resection piece and its concordant response rate.

ELIGIBILITY:
Inclusion Criteria:

* patients with DHG on Barrett's esophagus on endoscopic biopsies followed by endoscopic resection.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with DHG on Barrett's esophagus on endoscopic biopsies followed by endoscopic resection.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Influence of histological concordance on the risk of recurrence | 1 day
  the histological concordance being the comparison between the biopsies and the endoscopic resection piece and its concordant response rate.

SECONDARY OUTCOMES:
Identification of histological factors of recurrence. | 1 day
  Identification of histological factors of recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli-Calmettes, Marseille, Bouches-du Rhône, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Godat S, Caillol F, Autret A, Bories E, Pesenti C, Ratone JP, De Cassan C, Poizat F, Giovannini M. Endotherapy in case of relapse of neoplastic Barrett's esophagus after successful initial endoscopic resection. Surg Endosc. 2017 Sep;31(9):3703-3710. doi: 10.1007/s00464-016-5409-5. Epub 2017 Jan 11. PMID 28078459